CLINICAL TRIAL: NCT07221864
Title: Decoding Emotional Dynamics Driving Mood Instability in Bipolar Disorder
Brief Title: Decoding Emotional Dynamics in Bipolar Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Masaya Misaki, Associate Investigator, Laureate Institute for Brain Research, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-005; 5P20GM121312-08 (NIH)
Record Dates: First submitted 2025-10-23; First posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Bipolar Disorder I or II; Healthy (Controls)
Keywords: neuroimaging; fMRI; Bipolar Disorder I; Bipolar Disorder II; machine learning; emotion regulation
MeSH Terms: conditions — Bipolar Disorder; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decoding Emotional Dynamics (Experimental): All participants complete the same two-session protocol: a preparation visit with diagnostic interviews and questionnaires, followed by an MRI session including resting-state and task-based scans. During the Think and Regulate Affective States Task (TReAT), participants recall personal positive and negative memories, rate their emotions, and practice positive emotion amplification strategies. Physiological signals are recorded throughout. Both individuals with bipolar disorder and healthy controls complete identical procedures for comparison of brain and emotional dynamics.
  Interventions: Behavioral: Think and Regulate Affective State Task

INTERVENTIONS:
Behavioral: Think and Regulate Affective State Task — Participants complete the Think and Regulate Affective States Task (TReAT) during fMRI scanning. This task presents brief cues of participants' own autobiographical memories, four positive and four negative, to evoke corresponding emotional states. While viewing these cues, participants alternate between thinking about the memory, rating emotional valence and arousal, and practicing positive emotion amplification strategies. Each session includes multiple blocks of "Think," "Rate," "Regulate," "Attention," and "Rest" periods. Physiological measures (heart rate and respiration) are recorded concurrently. The task is designed to decode emotional states from fMRI data and evaluate the neural impact of positive emotion regulation in bipolar disorder compared to healthy controls.

SUMMARY:
The goal of this neuroimaging study is to investigate how emotional states fluctuate in people with bipolar disorder (BD) compared to healthy controls, and to understand the neural mechanisms driving mood instability. The main questions it aims to answer are:

* Can emotional states be decoded from fMRI brain activity using machine learning?
* Do individuals with BD show more unstable emotional state trajectories (e.g., high metastability, low fractal scaling) than healthy controls?
* Does amplifying positive emotions stabilize brain and emotional dynamics in BD?

Researchers will compare individuals with bipolar disorder (BD-I or BD-II, currently depressed or mixed state) to healthy controls without psychiatric history to see whether the BD group shows greater fluctuations in emotional brain activity and whether positive emotion regulation strategies normalize this instability.

Participants will:

* Complete self-report questionnaires on mood, emotion regulation, anxiety, and daily functioning.
* Recall and provide short descriptions of personal positive and negative memories to be used in the MRI task.
* Undergo fMRI scanning, including:
* Resting-state scans
* A Think and Regulate Affective States Task (TReAT) where they recall autobiographical memories, rate emotions, and practice amplifying positive mood.
* Structural and diffusion MRI for brain mapping.
* Receive physiological monitoring (heart rate, respiration) during scanning.
* Complete post-scan surveys on emotional state and task experience.

This research will help clarify how the brain supports or disrupts emotional regulation in bipolar disorder and may inform the development of personalized, neurobiologically informed treatments for mood instability.

DETAILED DESCRIPTION:
This neuroimaging study investigates the neural mechanisms underlying emotional dynamics and mood instability in individuals with bipolar disorder (BD). Bipolar disorder is characterized by rapid and intense mood fluctuations, yet the neurobiological basis of these transitions, how the brain shifts between emotional states in real time, remains poorly understood. The study aims to identify the moment-to-moment brain processes that drive emotional lability and to explore whether positive emotion amplification can stabilize emotional and neural states in BD.

Study Design

This is a study conducted at the Laureate Institute for Brain Research (LIBR) in Tulsa, Oklahoma. The study includes 72 participants total: 36 adults diagnosed with bipolar disorder type I or II (currently in a depressive or mixed state) and 36 healthy control participants without psychiatric history. Participants will complete two visits:

* A preparation session for consent, clinical interviews, and questionnaire completion, and
* A MRI scanning session that includes both resting-state and task-based fMRI.

Data will be collected using multimodal methods, including functional magnetic resonance imaging (fMRI), diffusion weighted imaging (DWI), structural MRI, and physiological monitoring (heart rate, respiration). Behavioral and emotional measures will be recorded throughout the study to align neural data with subjective emotional experience.

Scientific Rationale Mood instability is a defining and impairing feature of bipolar disorder, associated with deficits in emotion regulation and cognitive control. Prior neuroimaging work has identified alterations in prefrontal-limbic circuitry, including decreased activation in regulatory regions such as the anterior cingulate cortex (ACC) and prefrontal cortex (PFC), and increased activation in emotion-responsive regions such as the amygdala. However, most studies examine static mood states rather than dynamic fluctuations in emotional experience.

The present study applies machine learning, complexity science, and network control theory to quantify and model emotional state dynamics. By decoding brain activity during emotion regulation tasks, the research aims to characterize how emotional states evolve over time, how this differs in BD compared to healthy controls, and whether targeted regulation strategies, specifically positive emotion amplification, can modulate these dynamics.

Specific Aims and Hypotheses Aim 1: Decode momentary emotional states from whole-brain fMRI data using machine learning approaches.

Hypothesis 1: A machine learning classifier can accurately distinguish distinct emotional states (e.g., rumination vs. positive reflection) from fMRI activation patterns. BD participants will exhibit more unstable, fluctuating state trajectories than healthy controls.

Aim 2: Quantify emotional dynamics using metrics from complexity science and network control theory.

Hypothesis 2: Individuals with BD will show higher emotional metastability and lower fractal scaling-indicators of greater temporal irregularity in brain activity-relative to healthy controls. Network control theory analysis will identify the brain regions that contribute to state transitions.

Aim 3: Examine the effects of positive emotion amplification on emotional stability and brain network dynamics.

Hypothesis 3: The regulation of positive affect will engage cognitive control regions (e.g., dorsolateral PFC, ACC) and promote more stable emotional trajectories in BD participants.

Experimental Tasks and Procedures

* Visit 1 (Preparation Session):

Participants will undergo informed consent, psychiatric screening (using the MINI), and a series of standardized questionnaires assessing mood, emotion regulation, anxiety, rumination, and hedonic capacity (e.g., MADRS, YMRS, PANAS-X, DERS, ERQ, STAI, PROMIS scales).

Participants will also recall eight autobiographical events-four positive (reminiscence) and four negative (rumination)-and write brief keyword descriptions of each. These personalized cues will be used later in the MRI task to elicit emotional states without revealing personal content.

* Visit 2 (MRI Scanning Session):

Participants will complete both resting-state and task-based MRI scans lasting up to two hours. Physiological signals (heart rate and respiration) will be recorded concurrently to remove physiological artifacts and examine autonomic correlates of emotion.

MRI sequences include:

* High-resolution T1-weighted structural scans
* Diffusion-weighted scans for white-matter connectivity
* Resting-state fMRI (12-minute duration)
* Task fMRI: Think and Regulate Affective States Task (TReAT)

TReAT Task Overview

The Think and Regulate Affective States Task (TReAT) is a novel paradigm designed to model real-world emotional processing. Participants are presented with brief cue words corresponding to their personal autobiographical events and alternate between several types of blocks:

* Think Blocks: Participants think about the cued event, immersing themselves in the associated emotional experience.
* Rating Blocks: Immediately after, they rate emotional valence (positive-negative) and arousal using the Affective Slider.
* Regulation Blocks: Participants attempt to amplify positive mood while focusing on the same cue.
* Attention Blocks: Participants perform a brief arrow-direction attention task (6 trials, 2 seconds each) to clear cognitive load between emotional blocks.
* Rest Blocks: Participants fixate on a cross, instructed to relax and clear their thoughts.

These blocks are repeated across four fMRI runs, each lasting approximately 12-15 minutes. The design allows modeling of both spontaneous and regulated emotional states, enabling fine-grained temporal decoding of emotional dynamics.

After each run, participants rate fatigue, sleepiness, and emotional engagement. Post-scan questionnaires (e.g., PANAS-X, STAI-S, Feedback Questionnaire) assess emotional and physical comfort.

Data Analysis Plan Functional MRI data will be preprocessed using standard pipelines and analyzed with multivariate pattern analysis (MVPA) to classify emotional states. State-space trajectory analyses will examine how decoded brain states fluctuate over time within and between subjects. Measures of metastability, fractal scaling, and network controllability will quantify the temporal complexity and flexibility of brain networks.

Between-group comparisons (BD vs. HC) will assess whether BD participants exhibit greater temporal irregularity or reduced control energy in emotion-related circuits. The modulation of these parameters by positive emotion regulation will be tested using within-subject contrasts of Regulation vs. Think blocks.

Scientific and Clinical Significance This study integrates cutting-edge computational methods: machine learning, complexity metrics, and network control theory to decode the temporal structure of emotion regulation in bipolar disorder. By identifying neurobiological signatures of instability and testing whether positive affect regulation stabilizes these dynamics, this work aims to bridge the gap between affective neuroscience and personalized psychiatry.

The resulting dataset will contribute to the National Institute of Mental Health (NIMH) Data Archive and inform future large-scale studies targeting biomarkers of emotional dysregulation. Ultimately, this research will lay the groundwork for adaptive, brain-state-driven treatments that dynamically respond to patients' emotional states, offering new strategies for mood stabilization in bipolar disorder.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 to 65 years
2. Male or female
3. BMI between 18.5 and 38.0 kg/m2 at Screening
4. Capable of understanding and complying with study requirements
5. Fluent in English
6. Able to provide informed consent

   BD Group:
7. Meet the DSM-5 diagnostic criteria for BD-I or BD-II who are currently depressed or mixed state defined by the Mini-International Neuropsychiatric Interview (MINI)
8. Moderate or greater depressive symptom severity (MADRS ≥ 15 or PHQ-9 ≥ 10)

   HC Group:
9. No current or past psychiatric disorder (verified by MINI)

Exclusion Criteria

1. No telephone or easy access to a telephone
2. Significant medical problems as identified by the medical screening questionnaire: e.g. a history of unstable liver or renal insufficiency; glaucoma; significant and unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disturbance; or any other condition that, in the opinion of the investigator, would make participation not be in the best interest (e.g., compromise the well-being) of the participant or that could prevent, limit, or confound the protocol-specified assessments
3. A positive test for drugs of abuse, including alcohol (breath test), cocaine, opiates, amphetamines, methamphetamines, phencyclidine, benzodiazepines, barbiturates, methadone, and oxycodone
4. Drug or alcohol intoxication (based on positive UTOX or breathalyzer test at screening or study session) or reported alcohol/drug withdrawal, last cannabis use must be >48 hours prior to study session.
5. Current DSM-5 diagnosis of a psychosis spectrum disorder or moderate to severe substance use disorder
6. Moderate to severe traumatic brain injury or other neurocognitive disorder with evidence of neurological deficits, neurological disorders, or severe or unstable medical conditions that might be compromised by participation in the study (to be determined by primary care provider)
7. Current significant suicidal ideation or suicide attempt within the past 3 months.
8. Change in the dose or prescription of a medication within the 6 weeks before enrolling in the study that could affect brain functioning, e.g., anxiolytics, antipsychotics, antidepressants, or mood stabilizers
9. Taking drugs that affect the fMRI hemodynamic response (e.g., methylphenidate, acetazolamide, excessive caffeine intake > 1000 mg/day)
10. MRI contraindications as documented on the MR Environment Screening
11. Unwillingness or inability to complete any of the major aspects of the study protocol, including magnetic resonance imaging (i.e., due to claustrophobia), or behavioral assessment. However, failing to complete some individual aspects of these assessment sessions will be acceptable (i.e., being unwilling to answer individual items on some questionnaires or being unwilling to complete a behavioral task)
12. Non-correctable vision or hearing problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Decoded Emotional State Trajectory | Day 2
  The decoded emotional state time course derived from fMRI during the Think and Regulate Affective States Task (TReAT). Temporal irregularity will be quantified using permutation entropy to assess emotional state instability in individuals with bipolar disorder compared to healthy controls.
Metastability of brain network states | Day 2
  Metastability of brain network states will be calculated from whole-brain fMRI data to characterize variability in emotional states.

SECONDARY OUTCOMES:
Brain regional contributions to the transition energy of emotional brain state changes | Day 2
  Brain regional contributions to the transition energy of emotional brain state changes, derived from network control theory, will be calculated to identify regions that drive transitions between emotional states.
Fractal scaling of brain state changes | Day 2
  Fractal scaling of brain state changes will be calculated from whole-brain fMRI data to characterize the regularity of emotional brain states.

CONTACTS AND LOCATIONS:
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) from this study may be shared through public research repositories such as the National Institute of Mental Health (NIMH) Data Archive (NDA) following study completion. Shared data may include de-identified participant demographics, behavioral and questionnaire responses, functional and structural neuroimaging data, and study participation details. Data will be stripped of all identifying information in compliance with HIPAA and institutional standards for de-identification.
  To enable data sharing, information required to generate a Global Unique Identifier (GUID) will be collected according to NDA specifications. All data will be stored securely on encrypted servers and retained for at least three years after study completion, in accordance with federal and institutional requirements.
  Study findings will be disseminated through peer-reviewed journal publications, scientific conferences, and public data repositories.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Access Criteria: Qualified researchers with approved data use agreements may request access through the National Institute of Mental Health (NIMH) Data Archive (NDA). Access requires institutional affiliation, completion of the NDA Data Use Certification process, and agreement to comply with all confidentiality, security, and ethical use requirements. Data will be shared only in de-identified form through the NDA's secure access system; no direct identifiers or contact information will be provided.

REFERENCES:
- [Background] Betella A, Verschure PF. The Affective Slider: A Digital Self-Assessment Scale for the Measurement of Human Emotions. PLoS One. 2016 Feb 5;11(2):e0148037. doi: 10.1371/journal.pone.0148037. eCollection 2016. PMID 26849361
- [Background] Jubran A. Pulse oximetry. Crit Care. 2015 Jul 16;19(1):272. doi: 10.1186/s13054-015-0984-8. PMID 26179876
- [Background] Kryza-Lacombe M, Pearson N, Lyubomirsky S, Stein MB, Wiggins JL, Taylor CT. Changes in neural reward processing following Amplification of Positivity treatment for depression and anxiety: Preliminary findings from a randomized waitlist controlled trial. Behav Res Ther. 2021 Jul;142:103860. doi: 10.1016/j.brat.2021.103860. Epub 2021 Apr 15. PMID 33894554
- [Background] Nolen-Hoeksema S, Morrow J. A prospective study of depression and posttraumatic stress symptoms after a natural disaster: the 1989 Loma Prieta Earthquake. J Pers Soc Psychol. 1991 Jul;61(1):115-21. doi: 10.1037//0022-3514.61.1.115. PMID 1890582
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Misaki M, Phillips R, Zotev V, Wong CK, Wurfel BE, Krueger F, Feldner M, Bodurka J. Brain activity mediators of PTSD symptom reduction during real-time fMRI amygdala neurofeedback emotional training. Neuroimage Clin. 2019;24:102047. doi: 10.1016/j.nicl.2019.102047. Epub 2019 Oct 22. PMID 31711031
- [Background] Taylor CT, Lyubomirsky S, Stein MB. Upregulating the positive affect system in anxiety and depression: Outcomes of a positive activity intervention. Depress Anxiety. 2017 Mar;34(3):267-280. doi: 10.1002/da.22593. Epub 2017 Jan 6. PMID 28060463
- [Background] Hancock F, Cabral J, Luppi AI, Rosas FE, Mediano PAM, Dipasquale O, Turkheimer FE. Metastability, fractal scaling, and synergistic information processing: What phase relationships reveal about intrinsic brain activity. Neuroimage. 2022 Oct 1;259:119433. doi: 10.1016/j.neuroimage.2022.119433. Epub 2022 Jul 1. PMID 35781077
- [Background] Gu S, Pasqualetti F, Cieslak M, Telesford QK, Yu AB, Kahn AE, Medaglia JD, Vettel JM, Miller MB, Grafton ST, Bassett DS. Controllability of structural brain networks. Nat Commun. 2015 Oct 1;6:8414. doi: 10.1038/ncomms9414. PMID 26423222
- [Background] Misaki, M., et al. Decoding Temporal Dynamics of Emotion Regulation: Reinterpretation, Distraction, and Mindfulness. in OHBM 2025 - Annual Meeting Organization for Human Brain Mapping. 2025. Brisbane, Australia.
- [Background] Du M, Zhang L, Li L, Ji E, Han X, Huang G, Liang Z, Shi L, Yang H, Zhang Z. Abnormal transitions of dynamic functional connectivity states in bipolar disorder: A whole-brain resting-state fMRI study. J Affect Disord. 2021 Jun 15;289:7-15. doi: 10.1016/j.jad.2021.04.005. Epub 2021 Apr 20. PMID 33906006
- [Background] Han KM, De Berardis D, Fornaro M, Kim YK. Differentiating between bipolar and unipolar depression in functional and structural MRI studies. Prog Neuropsychopharmacol Biol Psychiatry. 2019 Apr 20;91:20-27. doi: 10.1016/j.pnpbp.2018.03.022. Epub 2018 Mar 28. PMID 29601896
- [Background] Houenou J, Frommberger J, Carde S, Glasbrenner M, Diener C, Leboyer M, Wessa M. Neuroimaging-based markers of bipolar disorder: evidence from two meta-analyses. J Affect Disord. 2011 Aug;132(3):344-55. doi: 10.1016/j.jad.2011.03.016. Epub 2011 Apr 5. PMID 21470688
- [Background] Janiri D, Frangou S. Precision neuroimaging biomarkers for bipolar disorder. Int Rev Psychiatry. 2022 Nov-Dec;34(7-8):727-735. doi: 10.1080/09540261.2022.2106121. Epub 2022 Aug 30. PMID 36786111
- [Background] Gruber J, Purcell AL, Perna MJ, Mikels JA. Letting go of the bad: deficit in maintaining negative, but not positive, emotion in bipolar disorder. Emotion. 2013 Feb;13(1):168-75. doi: 10.1037/a0029381. Epub 2012 Aug 6. PMID 22866884
- [Background] Ortiz A, Alda M. The perils of being too stable: mood regulation in bipolar disorder. J Psychiatry Neurosci. 2018 Nov 1;43(6):363-365. doi: 10.1503/jpn.180183. No abstract available. PMID 30371048

DOCUMENTS (2):
  • Study Protocol (2025-10-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT07221864/Prot_000.pdf
  • Informed Consent Form (2025-06-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT07221864/ICF_001.pdf